CLINICAL TRIAL: NCT04005846
Title: Transcranial Direct Current Stimulation (tDCS) to Improve Maximal Aerobic Performance in Recreational and Trained Runners
Brief Title: tDCS to Increase Aerobic Performance in Runners
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Géraldine Martens, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CE2019/186
Record Dates: First submitted 2019-06-21; First posted 2019-07-02 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Athletic Performance
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind randomized sham controlled crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS first / Sham tDCS second (Other): Receiving active tDCS during the first visit followed by sham tDCS on the next visit
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS first / Active tDCS second (Other): Receiving sham tDCS during the first visit followed by active tDCS on the next visit
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — The active session of tDCS will consist in applying two anodes over M1 bilaterally (C3 and C4 according to the 10-20 international EEG placement) and the cathodes over the occipital areas (O1 and O2), and to inject 2 mA for 20 minutes through sponge electrodes (35 cm²) placed on the scalp using the Startsim 8 (Neuroelectrics, Barcelona). The sham tDCS will use the same montage and device but direct current will only be injected for 30 seconds, with a ramp-up and ramp-down 15 seconds period, to mimic the somatosensory effects of active tDCS.

SUMMARY:
Many different factors affect running performance, transcranial direct current stimulation (tDCS) is a widely used and available neuromodulation tool and could hypothetically facilitate the supraspinal drive and thereby act upstream of the motor cortex to prolong the muscles work in time to exhaustion trials. While it appears to decrease the rating of perceived exertion (RPE) during cycling, little is known about the effects of tDCS on physiological performance parameters such as maximal oxygen consumption (VO2max), maximal aerobic speed (MAS) and lactate thresholds in runners.

The aim of this prospective randomized sham-controlled clinical trial is to investigate the physiological effects of tDCS applied over the motor cortex on perceived exertion and performance-related parameters measured by an incremental treadmill test to exhaustion.

This research thus aims at answering the following questions:

1. Is active tDCS applied bilaterally over the motor cortex significantly more efficient than sham tDCS to improve the TTE?
2. Does active tDCS decreases the RPE, as compared to sham?
3. Is there any significant difference between active and sham tDCS on the physiological parameters measured during an incremental test to exhaustion, namely: VO2max, MAS, respiratory exchange ratio, blood lactate levels, maximal heart rate?
4. Does the baseline level of physical fitness influences response to tDCS?

The investigators hypothesize that 1) performance as measured by time to exertion will be increased following active and not sham tDCS due to a decreased perceived rate of exertion without significantly altering the other physiological parameters; and 2) performance as measured by incremental treadmill test to exhaustion will be more improved in recreational as compared to trained runners.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Regular running activity above 2 hours/week
* VO2max above 30 mL/min/kg

Exclusion Criteria:

* Pacemaker
* Intracerebral metallic implant
* Smoking
* Using dietary supplementation or medication potentially affecting the CNS
* Musculoskeletal injury within the past 6 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Time to exertion (active vs. sham) | Immediate
  Time to achieve exhaustion during a treadmill test where the speed is set at a constant 90% of the individual maximal aerobic speed (determined during the screening visit)

SECONDARY OUTCOMES:
Ratings of perceived exertion (RPE) evolution (active vs. sham) | Every 3 minutes during the test to exhaustion until the end of the test (up to 1 hour after the stimulation)
  RPE will be assessed continuously (every 3 minutes) during the time to exhaustion trial using the Borg rating of perceived exertion scale (RPE scale). The Borg RPE scale is a quantitative measure of perceived exertion during physical activity. The scale starts with "no feeling of exertion," which rates a 6, and ends with "very, very hard," which rates a 20. Moderate activities register 11 to 14 on the Borg scale ("fairly light" to "somewhat hard"), while vigorous activities usually rate a 15 or higher ("hard" to "very, very hard").
Maximal Oxygen Consumption (VO2max) evolution (active vs. sham) | Immediate
  VO2max will be assessed continuously during the time to exhaustion trial using a gas analyzer
Lactate thresholds (active vs. sham) | Every 3 minutes during the test to exhaustion until the end of the test (up to 1 hour after the stimulation)
  Levels of blood lactate will be measured continuously (every 3 minutes) during the time to exhaustion trial using capillary blood and a lactate analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- ISEPK ULiège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martens G, Hody S, Bornheim S, Angius L, De Beaumont L, Fregni F, Ruffini G, Kaux JF, Thibaut A, Bury T. Can transcranial direct current stimulation (tDCS) over the motor cortex increase endurance running performance? a randomized crossover-controlled trial. PLoS One. 2024 Dec 5;19(12):e0312084. doi: 10.1371/journal.pone.0312084. eCollection 2024. PMID 39637186